CLINICAL TRIAL: NCT02943694
Title: The Feasibility and Safety of Instruments in Transanal Total Mesorectal Excision (TaTME) for Rectal Cancer
Acronym: FSI-TaTME
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Weiguo Hu, Vice President, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FT-001
Record Dates: First submitted 2016-10-20; First posted 2016-10-25 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Postoperative Complications
Keywords: TaTME; Complications; Instrument
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TaTME with CS-Compact (GelPoint Path) (Experimental): Based on newly-designed devices tailored for transanal TME, CS-Compact, GelPoint and Octoport are employed for the clinical applications.
  Interventions: Device: TaTME with CS-Compact (GelPoint pathway)

INTERVENTIONS:
Device: TaTME with CS-Compact (GelPoint pathway) — Standard TaTME with circular stapler (Short and straight, CS Compact), designed for extra-corporeal and endo-anal anastomosis procedures.

SUMMARY:
Colorectal cancer is one of the leading deadly diseases in the world. Due to the TME (total mesorectal excision) for the last decades, the survival and relapse rate of rectal cancer patients have been considerably improved. However, anatomical limitations in pelvic space hinder the further optimization of surgical treatment Thus, the natural orifice transluminal endoscopic surgery (NOTES) emerges as an alternative surgical strategy. Of note, transanal total mesorectal excision (TaTME) , a new invention based on TME principle, NOTES conception and single port technique, has been prevailing both in West and East nations, with or without the abdominal laparoscopic assistance. Up to date, there are various kinds of instruments and patterns to complete TaTME with comparable clinical outcomes. However, flaws in each instrument remains according to the feedbacks. This study is therefore designed to clinically evaluate the feasibility and safety of the new instruments specifically for TaTME (CS-Compact, GelPoint pathway).

DETAILED DESCRIPTION:
Rectal cancer comprises the most in colorectal cancer around the world, among which surgery remains the optimal therapeutic intervention. The TME (Total Mesorectal Excision), proposed by Bill Heald, provides novel insights for the eradication of possible disseminated cancer cells and therefore reduces the recurrence and mortality rates. However, either laparoscopic or open TME surgery is limited by the pelvic space and further improvement. For the last decade, the emerging of the natural orifice transluminal endoscopic surgery (NOTES) offers an alternative pattern for rectal cancer surgery, among which, the TaTME (transanal total mesorectal excision) represents the most optimized surgery techniques. Derived from TME, NOTES and modified laparoscopic instruments, TaTME facilitates the dissection process of rectal cancer from caudal to cranial, from indirect to direct vision. TaTME allows for accurate confirmation of resected margin with proper transecting level, better dissection of mesorectum and protection of sphincter, a qualified end-to-end anastomosis and reduced need of endolinear stapler and possible leakage afterwards. However, various kinds of instruments and surgical procedures have been proposed to complete TaTME, all of which have been validated by preclinical and clinical trials in small size. Of note, this study is initiated to apply a suit of instruments specifically designed for TaTME ( GelPoint pathway CS-Compact) and clinically evaluate the feasibility and safety of the new instruments without comparison to other prevailing ones. The CS-Compact and GelPoint pathway has been confirmed both safe and feasible to operate in preclinical trials and clinical trials in western. This study strictly examines the corresponding issues in Chinese rectal cancer patients. The surgeons in our institute have successfully completed the training programs of TaTME in preclinical trials, in animal models and cadavers. Clinical skills and knowledge to safe operations are qualified.

ELIGIBILITY:
Inclusion Criteria:

* rectal cancer patients, confirmed by the endoscopic biopsy;
* curative rectal cancer in clinical stage with resectable lesion, the cTNM stage <T3 stage, with comparable tumor size in low or medial rectum.
* patients' general information, 18ys<age<75ys, no restriction in genders, BMI< or =30kg/m2, no presentation of severe chronic diseases (i.e. COPD), WHO classification <2 (Zubrod-ECOG-WHO)
* patients or representatives have agreed and signed the informed consent documents.

Exclusion Criteria:

* have received neo-adjuvant chemotherapy or radiotherapy before operations;
* previous surgery in pelvis
* uncontrollable diseases such as diseases in cardiopulmonary function, chronic bronchitis, severe hepatitis/diabetes/malnutrition/renal function.
* suffer from other malignant diseases, i.e. gastric cancer, liver cancer.
* pregnant, lactation stage.
* metal disorders.
* lacking qualified compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with post-operative complications | postoperative 30days (hospital-stay time course)
  Number of participants with post-operative complications (e.g. numbers of postoperative bleeding, leakage, infections)

SECONDARY OUTCOMES:
3-year disease free survival rate | postoperative 3years
  3-year disease free survival rate （the period after curative treatment without any detection of disease ）, the detailed information of 3y-DFS will be obtained by period follow-up of patients by calls and outpatient checking.
3-year overall survival rate | postoperative 3years
  3-year overall survival rate （the survival period after curative treatment ）, the detailed information of 3y-OS will be obtained by period follow-up of patients by calls and outpatient checking.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Guo HU, Ph.D., M.D., Study Director — Ruijin Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Siegel R, Desantis C, Jemal A. Colorectal cancer statistics, 2014. CA Cancer J Clin. 2014 Mar-Apr;64(2):104-17. doi: 10.3322/caac.21220. Epub 2014 Mar 17. PMID 24639052
- [Background] Brenner H, Kloor M, Pox CP. Colorectal cancer. Lancet. 2014 Apr 26;383(9927):1490-1502. doi: 10.1016/S0140-6736(13)61649-9. Epub 2013 Nov 11. PMID 24225001
- [Background] Heald RJ, Ryall RD. Recurrence and survival after total mesorectal excision for rectal cancer. Lancet. 1986 Jun 28;1(8496):1479-82. doi: 10.1016/s0140-6736(86)91510-2. PMID 2425199
- [Background] MacFarlane JK, Ryall RD, Heald RJ. Mesorectal excision for rectal cancer. Lancet. 1993 Feb 20;341(8843):457-60. doi: 10.1016/0140-6736(93)90207-w. PMID 8094488
- [Background] McLemore EC, Harnsberger CR, Broderick RC, Leland H, Sylla P, Coker AM, Fuchs HF, Jacobsen GR, Sandler B, Attaluri V, Tsay AT, Wexner SD, Talamini MA, Horgan S. Transanal total mesorectal excision (taTME) for rectal cancer: a training pathway. Surg Endosc. 2016 Sep;30(9):4130-5. doi: 10.1007/s00464-015-4680-1. Epub 2015 Dec 10. PMID 26659246
- [Background] Telem DA, Han KS, Kim MC, Ajari I, Sohn DK, Woods K, Kapur V, Sbeih MA, Perretta S, Rattner DW, Sylla P. Transanal rectosigmoid resection via natural orifice translumenal endoscopic surgery (NOTES) with total mesorectal excision in a large human cadaver series. Surg Endosc. 2013 Jan;27(1):74-80. doi: 10.1007/s00464-012-2409-y. Epub 2012 Jun 30. PMID 22752277
- [Background] Atallah S, Albert M, Larach S. Transanal minimally invasive surgery: a giant leap forward. Surg Endosc. 2010 Sep;24(9):2200-5. doi: 10.1007/s00464-010-0927-z. Epub 2010 Feb 21. PMID 20174935
- [Background] Kneist W, Hanke L, Kauff DW, Lang H. Surgeons' assessment of internal anal sphincter nerve supply during TaTME - inbetween expectations and reality. Minim Invasive Ther Allied Technol. 2016 Oct;25(5):241-6. doi: 10.1080/13645706.2016.1197269. Epub 2016 Jun 22. PMID 27333465
- [Background] Muratore A, Mellano A, Marsanic P, De Simone M. Transanal total mesorectal excision (taTME) for cancer located in the lower rectum: short- and mid-term results. Eur J Surg Oncol. 2015 Apr;41(4):478-83. doi: 10.1016/j.ejso.2015.01.009. Epub 2015 Jan 17. PMID 25633642